CLINICAL TRIAL: NCT03762148
Title: The Effect of Prebiotics on Iron Absorption in Women With Low Iron Stores: Determination of a Dose-dependent Effect of Galacto-oligosaccharides on Iron Absorption, With and Without Addition of Ascorbic Acid
Brief Title: Determination of a Dose-dependent Effect of GOS on Iron Absorption, and Addition of Vitamin C
Acronym: Fe_GOS_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Burgerstein Vitamine (Industry)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, PhD, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Fe_GOS_2
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Iron-deficiency
Keywords: iron-deficiency; prebiotics; galacto-oligosaccharides
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate; ferrous sulfate; ferric pyrophosphate; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- ferrous fumarate (Experimental): labelled iron as ferrous fumarate
  Interventions: Dietary Supplement: ferrous fumarate
- ferrous sulphate (Experimental): labelled iron as ferrous sulphate
  Interventions: Dietary Supplement: ferrous sulphate
- ferric pyrophosphate (Experimental): labelled iron as ferric pyrophosphate
  Interventions: Dietary Supplement: ferric pyrophosphate
- ferrous fumarate + 3.5 g GOS (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 3.5 g GOS
  Interventions: Dietary Supplement: ferrous fumarate + 3.5 g GOS
- ferrous fumarate + 7 g GOS (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 7 g GOS
  Interventions: Dietary Supplement: ferrous fumarate + 7 g GOS
- ferrous sulphate + 15 g GOS (Experimental): labelled iron as ferrous sulphate + prebiotics in the form of 15 g GOS
  Interventions: Dietary Supplement: ferrous sulphate + 15 g GOS
- ferrous fumarate + Vitamin C (Experimental): labelled iron as ferrous fumarate + Vitamin C
  Interventions: Dietary Supplement: ferrous fumarate + Vitamin C
- ferric pyrophosphate + 15 g GOS (Experimental): labelled iron as ferric pyrophosphate + prebiotics in the form of 15 g GOS
  Interventions: Dietary Supplement: ferric pyrophosphate + 15 g GOS
- ferrous fumarate + 7 g GOS + Vitamin C (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 7 g GOS + Vitamin C
  Interventions: Dietary Supplement: ferrous fumarate + 7 g GOS + Vitamin C

INTERVENTIONS:
Dietary Supplement: ferrous fumarate — nutritional iron (14 mg) supplement in form of ferrous fumarate
  Arms: ferrous fumarate
Dietary Supplement: ferrous sulphate — nutritional iron (14 mg) supplement in form of ferrous sulphate
  Arms: ferrous sulphate
Dietary Supplement: ferric pyrophosphate — nutritional iron (14 mg) supplement in form of ferric pyrophosphate
  Arms: ferric pyrophosphate
Dietary Supplement: ferrous fumarate + 3.5 g GOS — nutritional iron (14 mg) supplement in form of ferrous fumarate with addition of prebiotics (3.5 g GOS)
  Arms: ferrous fumarate + 3.5 g GOS
Dietary Supplement: ferrous fumarate + 7 g GOS — nutritional iron (14 mg) supplement in form of ferrous fumarate with addition of prebiotics (7 g GOS)
  Arms: ferrous fumarate + 7 g GOS
Dietary Supplement: ferrous sulphate + 15 g GOS — nutritional iron (14 mg) supplement in form of ferrous sulphate with addition of prebiotics (15 g GOS)
  Arms: ferrous sulphate + 15 g GOS
Dietary Supplement: ferrous fumarate + Vitamin C — nutritional iron (14 mg) supplement in form of ferrous fumarate with addition of Vitamin C
  Arms: ferrous fumarate + Vitamin C
Dietary Supplement: ferric pyrophosphate + 15 g GOS — nutritional iron (14 mg) supplement in form of ferric pyrophosphate with addition of prebiotics (15 g GOS)
  Arms: ferric pyrophosphate + 15 g GOS
Dietary Supplement: ferrous fumarate + 7 g GOS + Vitamin C — nutritional iron (14 mg) supplement in form of ferrous fumarate with addition of prebiotics (7 g GOS) and Vitamin C
  Arms: ferrous fumarate + 7 g GOS + Vitamin C

SUMMARY:
Iron deficiency is still the most common and widespread nutritional disorder in the world according to WHO.

In a recent iron absorption study in adult women with low iron stores in our lab (publication under review), we found that 15 g of GOS given with an iron supplement in the form of iron fumarate acutely increased iron absorption when given with water and a bread based meal. The dose of 15 g of GOS was tolerated well by the participants. As a follow up to the study mentioned above, we want to investigate: 1) if acute iron absorption is affected by lower doses of GOS; 2) whether this acute effect occurs for other commonly used iron compounds as well, such as iron sulphate and iron phosphate; and 3) if there are potential interactions on absorption with other enhancers of iron absorption, such as vitamin c.

DETAILED DESCRIPTION:
Iron is an important mineral in our body and fulfills essential functions such as for example oxygen transport from the lungs to the tissues. Iron deficiency is still the most common and widespread nutritional disorder in the world according to WHO. Common iron supplements all have their limitations in terms of availability and compatibility. Prebiotic fibers, such as galacto-oligosaccharides (GOS), selectively enhance growth of beneficial colonic bacteria. Prebiotics in general enhance the production of short-chain fatty acids (SCFAs) and thereby decrease luminal pH. Through the reduction in pH, prebiotics can enhance absorption of minerals such as calcium and magnesium and they have been proposed to potentially improve iron absorption.

In a recent iron absorption study in adult women with low iron stores in our lab (publication under review), we found that 15 g of GOS given with an iron supplement in the form of iron fumarate acutely increased iron absorption when given with water and a bread based meal. The dose of 15 g of GOS was tolerated well by the participants. As a follow up to the study mentioned above, we want to investigate: 1) if acute iron absorption is affected by lower doses of GOS; 2) whether this acute effect occurs for other commonly used iron compounds as well, such as iron sulphate and iron phosphate; and 3) if there are potential interactions on absorption with other enhancers of iron absorption, such as vitamin c.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* SF levels <30 µg/L
* Normal body Mass Index (18.5-24.9 kg/m2)
* Body weight <70 kg
* Signed informed consent

Exclusion Criteria:

* Severe anaemia (Hb < 80 g/L)
* Elevated CRP >10.0 mg/L
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole studies (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration, including pre- and-or probiotics supplements (excluding foods and beverages with life cultures such as yoghurt, raw milk cheese and kombucha)
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Difficulties with blood sampling
* Use of antibiotics over the past month
* Known hypersensitivity to iron supplements in the given amount, GOS, or lactose
* Women who are pregnant or breast feeding
* Women who intend become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, inject-able, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse -
* Smokers (> 1 cigarette per week)
* Inability to follow the procedures of the study, e.g. due to language problems, self-- reported psychological disorders, etc. of the participant
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are being studied
Enrollment: 46 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
fractional iron absorption | 2 months
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of several isotopically labelled iron supplements.Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, Dr., Principal Investigator — University of Zurich
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeroense FMD, Zeder C, Zimmermann MB, Herter-Aeberli I. Acute Consumption of Prebiotic Galacto-Oligosaccharides Increases Iron Absorption from Ferrous Fumarate, but not from Ferrous Sulfate and Ferric Pyrophosphate: Stable Iron Isotope Studies in Iron-Depleted Young Women. J Nutr. 2020 Sep 1;150(9):2391-2397. doi: 10.1093/jn/nxaa199. PMID 32692367